CLINICAL TRIAL: NCT04948138
Title: Glutamine Supplement in MELAS (Mitochondrial Encephalopathy, Lactic Acidosis, and Stroke-like Episodes) Syndrome in Order to Prevent Neurological Damage.
Brief Title: Glutamine Supplement in MELAS (Mitochondrial Encephalopathy, Lactic Acidosis, and Stroke-like Episodes) Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesús González de la Aleja Tejera (Other)
Responsible Party: Sponsor-Investigator, Jesús González de la Aleja Tejera, Jesús González de la Aleja Tejera, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLN-9-MIT
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: MELAS Syndrome
Keywords: MELAS; Glutamine; Oral supplements; Lactate; Cerebrospinal fluid; Magnetic resonance spectroscopy
MeSH Terms: conditions — MELAS Syndrome

STUDY DESIGN:
Intervention Model Description: Glutamine oral supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MELAS (Mitochondrial Encephalopathy, Lactic Acidosis, and Stroke-like episodes) syndrome (Experimental): Patients with MELAS syndrome that will receive oral supplementation with 10-15 g/day of glutamine (adjusted for weight and plasma concentrations)
  Interventions: Dietary Supplement: Glutamine oral supplementation

INTERVENTIONS:
Dietary Supplement: Glutamine oral supplementation — Oral supplementation with 10-15 g/day of glutamine (adjusted for weight and plasma concentrations).

SUMMARY:
The purpose of this study is to assesses the efficacy of oral supplementation with glutamine over three months on several amino acids and lactate concentration measured in cerebrospinal fluid and cerebral lactate measured by magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
Mitochondrial encephalomyopathy, lactic acidosis, and stroke-like episodes (MELAS) syndrome is a genetically heterogeneous disorder. The most common mutation is in the mtDNA gene MT-TL1 encoding the mitochondrial tRNALeu (UUR). For understanding the development of seizures in patients with mitochondrial disease, a study has recently emphasized the deficiency of astrocytic glutamine synthetase, creating a disinhibited neuronal network for seizure generation. The investigators propose to evaluate nine patients with mitochondrial DNA mutation and MELAS. Patients will receive oral supplementation with 10-15 g/day of glutamine (adjusted for weight and plasma concentrations). The primary outcome measures several amino acids (including glutamine) and lactate concentration measured in cerebrospinal fluid and cerebral lactate measured by magnetic resonance spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of MELAS syndrome is based on medical history (lactic acidosis, stroke-like episodes, and encephalomyopathy).
* Subjects have to be clinically stable for more than six months after any stroke-like episodes.
* All subjects have to be genetically confirmed.

Exclusion Criteria:

* Subjects harboring a MELAS-related pathogenic mtDNA mutation, no fulfilling the complete diagnostic criteria for the MELAS phenotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Amino Acids concentration in cerebrospinal fluid | 3 months
  Amino Acids (including glutamine) concentration measured in cerebrospinal fluid
Lactate concentration in cerebrospinal fluid | 3 months
  Lactate concentration measured in cerebrospinal fluid

SECONDARY OUTCOMES:
Lactate measured by magnetic resonance spectroscopy. | 3 months
  Cerebral Lactate measured by magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús González de la Aleja Tejera, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerrero-Molina MP, Bernabeu-Sanz A, Ramos-Gonzalez A, Morales-Conejo M, Delmiro A, Dominguez-Gonzalez C, Arenas J, Martin MA, Gonzalez de la Aleja J. Magnetic resonance spectroscopy in MELAS syndrome: correlation with CSF and plasma metabolite levels and change after glutamine supplementation. Neuroradiology. 2024 Mar;66(3):389-398. doi: 10.1007/s00234-023-03263-1. Epub 2023 Dec 19. PMID 38114794
- [Derived] Guerrero-Molina MP, Morales-Conejo M, Delmiro A, Moran M, Dominguez-Gonzalez C, Arranz-Canales E, Ramos-Gonzalez A, Arenas J, Martin MA, de la Aleja JG. High-dose oral glutamine supplementation reduces elevated glutamate levels in cerebrospinal fluid in patients with mitochondrial encephalomyopathy, lactic acidosis and stroke-like episodes syndrome. Eur J Neurol. 2023 Feb;30(2):538-547. doi: 10.1111/ene.15626. Epub 2022 Nov 18. PMID 36334048